CLINICAL TRIAL: NCT02866994
Title: Project Connect: Enhancing Connections During Metastatic Breast Cancer (PCO)
Brief Title: Project Connect Online: An Internet-based Intervention for Women With Breast Cancer
Acronym: PCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14-001744; 20155036 (Other Grant/Funding Number: Breast Cancer Research Foundation); SAC110009 (Other Grant/Funding Number: Susan G. Komen Breast Cancer Foundation)
Record Dates: First submitted 2016-08-01; First posted 2016-08-15 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-04

CONDITIONS: Breast Neoplasms
Keywords: Women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project Connect Online (PCO) (Experimental): Creation of personal website to share breast cancer experience with friends and family
  Interventions: Behavioral: Project Connect Online
- PCO PLUS (Experimental): Creation of personal website to share breast cancer experience with friends and family, as well as other women diagnosed with breast cancer
  Interventions: Behavioral: PCO PLUS

INTERVENTIONS:
Behavioral: Project Connect Online — Three-hour workshop to complete personal website regarding breast cancer experience to share with friends and family
  Arms: Project Connect Online (PCO)
Behavioral: PCO PLUS — Three-hour workshop to complete personal website regarding breast cancer experience to share with friends and family, as well as other women diagnosed with breast cancer
  Arms: PCO PLUS

SUMMARY:
This randomized comparative effectiveness trial examines the potential psychosocial and physical health-related benefits of sharing personal websites with other women with breast cancer, as well as with family and friends (PCO PLUS condition) versus sharing with family and friends only (PCO condition) in a sample of women with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* women at least 18 years of age;
* first diagnosis of Stage IV breast cancer or a recurrent diagnosis of metastatic breast cancer, any interval since diagnosis;
* ability to complete the intervention and assessments in English; and
* willingness to attend in-person PCO workshop;

Exclusion Criteria:

* male (because men constitute less than 1% of breast cancer patients, numbers would not be sufficient for reliable analyses);
* local (i.e., same breast, surgical scar, chest wall) or regional (i.e., lymph nodes) recurrent disease; and
* use of a personal website to post cancer-relevant material in the past six months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Change of general and cancer-related psychological status | Baseline, 2 months, 4 months
  web site self reported

SECONDARY OUTCOMES:
Change in overall physical health status | Baseline, 2 months, 4 months
  web site self reported

OTHER OUTCOMES:
Psychological mediator and moderator assessment | Baseline, 2 months, 4 months
  phone and web based assessment: Comparative effectiveness of the two conditions will be evaluated with analysis of covariance (ANCOVA), in which the dependent variable is CES-D (Center for Epidemiologic Studies-Depression scale, condition assignment and any variables on which baseline imbalance is observed.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Ganz, MD, Principal Investigator — Proffessor and Director, Health Policy & Management
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States